CLINICAL TRIAL: NCT02879461
Title: Prospective Study Comparing Surgical Decompression Associated With Physical Therapy And Physical Therapy Isolated In Patients With Lumbar Canal Stenosis
Brief Title: Surgical Decompression Associated With Physical Therapy and Physical Therapy Isolated in Patients With Lumbar Stenosis.
Acronym: Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Claudio Lacerda Rodrigues, Chief Of Orthopedics And Traumatology Discipline Medical School Santa Marcelina, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16127913.4.0000.5505
Record Dates: First submitted 2016-08-09; First posted 2016-08-25 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: LUMBAR STENOSIS
Keywords: SURGERY; REHABILITATION
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbar Decompression plus Physical Therapy (Active Comparator): First group will be submitted to lumbar decompression L3 to S1 and physical therapy with exercise Application of questionnaires Oswestry Rolland moris Sf 36 Of 6minutos walk test Likert scale Use of paracetamol
  Interventions: Procedure: LUMBAR DESCOMPRESSION
- Physical Therapy (Active Comparator): Second group physical therapy alone, with exercises Application of questionnaires Oswestry Rolland moris Sf 36 Of 6minutos walk test Likert scale Use of paracetamol
  Interventions: Procedure: LUMBAR DESCOMPRESSION

INTERVENTIONS:
Procedure: LUMBAR DESCOMPRESSION — ATRODESIS AND DESCOMPRESSIO OFF VERTEBRAL CANAL
  Other Names: LUMBAR STENOSIS

SUMMARY:
Stenosis of symptomatic lumbar canal is presented as a series of degenerative changes affecting the various vertebral segment structures, including: a joint zigoapofisária, yellow ligament, the articular capsule and the intervertebral disk. These changes decrease the area of the spinal canal and press the neural structures and may present clinically as the narrow tunnel syndrome.

This presentation was first described by Verbiest associated with these anatomical changes the clinical manifestations; corresponding to low back pain, pain in the legs that worsen with the fact ambulate and improve with rest, this presentation called neurogenic claudication .

The lumbar canal stenosis was divided into two main types; congenital and acquired . The first is associated with a reduced size of the pedicles, which leads to a reduction of the diameter of the spinal canal, common in patients achondroplasics . The acquired is considered the most common type and is associated with aging, including all anatomical structures of the lumbar segment .

With an aging population the number of symptomatic patients is increasing, although there is no statistic defined stenosis of symptomatic lumbar canal is the main reason for surgical approaches to the spine in patients over 60 years of age (7).

As described by Daffner et al a reduction in blood flow leads to production of inflammatory mediators, which associated with anatomical changes previously described lead to the clinical picture with lameness and pain in the lower limbs Treatment of these patients is beginning with guidance on the disease, adequate pain control, physical therapy and exercise for maintaining the activities of daily living. If these measures fail a surgical approach may be necessary, especially in patients with exercise intolerance, difficulty walking and urinary incontinence .

The surgical approach despite being widely studied in the literature prospective controlled studies are rare, found series of case studies or retrospective studies, we try to evaluate the effectiveness of surgery compared to rehabilitation in symptomatic patients in an attempt to assess the impact of surgery associated with comparing therapy with isolated therapy in these patients.

DETAILED DESCRIPTION:
Stenosis of symptomatic lumbar canal is presented as a series of degenerative changes affecting the various vertebral segment structures, including: a joint zigoapofisária, yellow ligament, the articular capsule and the intervertebral disk. These changes decrease the area of the spinal canal and press the neural structures and may present clinically as the narrow tunnel syndrome.

This presentation was first described by Verbiest associated with these anatomical changes the clinical manifestations; corresponding to low back pain, pain in the legs that worsen with the fact ambulate and improve with rest, this presentation called neurogenic claudication .

The lumbar canal stenosis was divided into two main types; congenital and acquired . The first is associated with a reduced size of the pedicles, which leads to a reduction of the diameter of the spinal canal, common in patients achondroplasics . The acquired is considered the most common type and is associated with aging, including all anatomical structures of the lumbar segment .

With an aging population the number of symptomatic patients is increasing, although there is no statistic defined stenosis of symptomatic lumbar canal is the main reason for surgical approaches to the spine in patients over 60 years of age .

As described by Daffner et al a reduction in blood flow leads to production of inflammatory mediators, which associated with anatomical changes previously described lead to the clinical picture with lameness and pain in the lower limbs Treatment of these patients is beginning with guidance on the disease, adequate pain control, physical therapy and exercise for maintaining the activities of daily living. If these measures fail a surgical approach may be necessary, especially in patients with exercise intolerance, difficulty walking and urinary incontinence .

The surgical approach despite being widely studied in the literature prospective controlled studies are rare, found series of case studies or retrospective studies, we try to evaluate the effectiveness of surgery compared to rehabilitation in symptomatic patients in an attempt to assess the impact of surgery associated with comparing therapy with isolated therapy in these patients.

2.OBJETIVOS The aim of this study is to evaluate the effectiveness of surgical approach associated with physiotherapy compared with physiotherapy alone in the quality of life in the lumbar narrow tunnel syndrome.

Secondary objectives: to evaluate the influence of physical therapy on muscle gain and improves the conditioning of these patients.

To evaluate the incidence of complications in patients undergoing surgical approach.

3. PATIENTS AND METHODS

3.1 - Delineation Our research contains a controlled prospective, randomized and blinded to the evaluator that evaluates the effectiveness of the surgical approach more physical therapy associated with isolated physical therapy in symptomatic lumbar spinal stenosis.

3.2 - Patients As research subjects will be randomized 62 patients through board electronic randomization ..

They will be included patients aged 50 to 75 years, of both genders, who agreed to participate in the work, having previously agreed to sign the consent form. Patients will be subject to an anthropometric assessment, with altitude record, weight and presence of associated comorbidities.

After the initial evaluation, patients will be randomized, with a group that will undergo surgery and after 3 weeks postoperatively initiated a rehabilitation program, a second group will be isolated physiotherapy. As an evaluation factor, also you will be given a bottle of paracetamol 750 mg and dated sheet, which will be instructed to register the day and the number of capsules taken for a period of 90 days.

3.3 - Clinical diagnosis In the clinical diagnosis of the case was the presence of claudication under walk 100m and at least two of the following complaints in lower limb pain, weakness, burning or tingling that worsens with walking and improves with the stop of ambulation and may or may not It is associated with low back pain.

3.4 - Radiological diagnosis In our study, the presence of lumbar canal stenosis was considered with an area less than 100mm2, based on criteria Hamanishi measured on MRI of the lumbar spine in follow-L3 to S1.

All patients underwent MRI on a device of 1 Tesla (Philips, Giroscan) belonging to the image of Hospital Santa Marcelina, SP. The test was done with the patient supine and cushion on his knees to maintain flexion of the hip and knee.

To avoid bias in the channel area due to the angle, all the cuts were made parallel to the discs, being accepted a difference of angle of at most 5.

The calculation was based on mathematical values, as follows: we calculated the laterolateral diameter (a) and anteroposterior (b) where the major axis whose data were provided by computer program (OSIRIX® 2010) on the scanned image. In case there were any differences, the figures would be recalculated and decided whether, then, for an average value between the measures. After calculating these values were divided by two, individually and multiplied by the value π (PI) . The obtained result is multiplied by a constant ranging from 0.8 (when the channel was circular), 0.7 (where the channel was elliptical), in the presence of 0.6 and 0.5 facet compression, when compression was made by the disc and the facets. Thus, (a / 2) x (b / 2) x π (constant) .

3.5 - Intervention

After the patient's initial assessment and the same take part in the study. Will be randomized in one of the groups the 1st group will be associated with decompression with arthrodesis implant placement type pedicle screws, are included patients requiring decompression of up to three levels. After three weeks of surgical treatment the patient started a rehabilitation program with physiotherapy assistance with weekly frequency for a period of 12 weeks.

The second group is subjected to a rehabilitation program isolated identical to the 1st group for 12 weeks.

Both groups will be offered 750 mg of paracetamol for up to 3 taken daily for 90 days. The evaluations will be carried out at the time of inclusion in the project, and the patient who undergoes surgery had performed surgery the following week after the assessment. The second evaluation will be conducted 4 weeks after, in both groups, this evaluation will be conducted to compare the muscle losses after surgery. The following evaluations will be performed in T12, 12 weeks after the start of rehabilitation, 24 and 48 weeks after the start of rehabilitation.

They will be also evaluated the incidence of complications in patients undergoing surgery.

Patients who are on medical treatment and opt for surgical treatment may do so at any time of the study.

As an auxiliary method of evaluation will be made a mensuramento the quadriceps diameter and sural triceps at all owner?.

3.6 - Assessment tools

1. Visual Analog Scale (VAS): instrument subjectively assesses the pain using a visual analog scale, in which the patient quantifies the degree of their pain following a line of 0 to 10 cm, with 0 being no pain and 10 unbearable pain (FERRAZ, 1990). The patient was asked about the pain he felt to walk last week.
2. Roland-Morris is extracted questionnaire physical component of the Sickness Impact Profile, plus in each question, the phrase "because of my back." This questionnaire consists of 24 questions relevant to the daily lives of individuals with low back pain, easy application, applied in less than 5 minutes and immediately score
3. 6-minute walk test: used to evaluate the functional capacity of the patient. The test was performed on a track of 22 meters traveled at a maximum speed achieved by the patient for six minutes following the guidelines of the American Thoracic Society (American Toracic Society (ATS) Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories).
4. Short Form SF36: generic instrument to assess quality of life, translated from English into Portuguese and validated with 36 questions divided into eight areas. In this questionnaire are discussed aspects related to functional capacity, limitations on physical aspects, pain, general health, vitality, social functioning, emotional aspects and mental health. The score ranges from zero to one hundred, zero being the worst health condition, and one hundred the best .
5. Scale Likert: It is a psychometric scale commonly used in questionnaires where the patient reports his opinion directly, according to their view of treatment: much better, somewhat better, not better, just worse and worse.
6. Disability Index Oswestry The ODI is used for functional evaluation of the lumbar spine, incorporating measures of pain and activity. The scale consists of 10 questions six alternatives, whose value ranges from 0 to 5.

3.7 - Calculation of n. Considering a 80% power and 5% significance, to compare VAS between the two groups at 5 different times, considering a standard deviation equal to 2 and a minimum difference between the measures equal to 2, it took 31 individuals in each group to greater certainty as to the validity of the results.

ELIGIBILITY:
Inclusion Criteria:

* claudication Presence less than 100m ambulation;
* Pain in the lower limbs;
* Weakness in lower limbs;
* Burning in the lower limbs;
* Tingling in the lower limbs;
* Low back pain;
* the lower spinal canal area to 100mm2, at the discretion of Hamanishi.

Exclusion Criteria:

* decompensated diabetes mellitus;
* Systemic hypertension and decompensated heart disease;
* Systemic diseases to occur in the lower limbs;
* Neuromuscular diseases;
* Patients with previous surgery in the lumbar or thoracic spine;
* Cognitive impairment that interferes with the ability to understand or interpret the questionnaires;

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Baseline, after 4, 12, 24 and 48 weeks
  Measured using the VAS

SECONDARY OUTCOMES:
Change in function | Baseline, after 4, 12, 24 and 48 weeks
  Measured using the Roland Morris questionnaire
Change in function | Baseline, after 4, 12, 24 and 48 weeks
  Measured using the Oswestry questionnaire
Change in walking distance | Baseline, after 4, 12, 24 and 48 weeks
  Measured using the six minute walking test
Change in quality of life | Baseline, after 4, 12, 24 and 48 weeks
  Measured using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Mareclina Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rodrigues LCL, Natour J. Surgical treatment for lumbar spinal stenosis: a single-blinded randomized controlled trial. Adv Rheumatol. 2021 May 12;61(1):25. doi: 10.1186/s42358-021-00184-6. PMID 33980309